CLINICAL TRIAL: NCT06184503
Title: A Real-world Analysis of Pharmacodynamic Response to Velmanase Alfa (Lamzede®) Treatment in Patients With Alpha-Mannosidosis Less Than 3 Years of Age
Brief Title: Analysis of Velmanase Alfa (Lamzede®)'s Effects in the Body of Children With Alpha-Mannosidosis Under the Age 3
Acronym: LAMPO(0-3)
Status: Recruiting | Type: Observational
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLI-LMZYMAA2-04
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Alpha-Mannosidosis
MeSH Terms: conditions — alpha-Mannosidosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paediatric patients with alpha-mannosidosis treated with Lamzede before 3 years of age: Paediatric patients with a confirmed diagnosis of alpha-mannosidosis with data for at least one pre- and one post-Lamzede treatment sample obtained when < 3 YOA.
  Interventions: Drug: Velmanase Alfa

INTERVENTIONS:
Drug: Velmanase Alfa — Lamzede® (velmanase alfa, henceforth referred to as Lamzede) is a recombinant human lysosomal alpha-mannosidase product developed as an intravenous enzyme replacement therapy (ERT) for the treatment of alpha-mannosidosis.
  Other Names: Lamzede

SUMMARY:
The goal of this observational study is to learn the effects of the drug velmanase alfa (Lamzede®) in the bodies of children under the age of 3 with Alpha-Mannosidosis.

The main questions it aims to answer are:

* study the effect of velmanase alfa on a marker of the disease called GlcNAc(Man)2 after one year of therapy
* explore how the child's body reacts to velmanase alfa during the therapy The parents or legal guardians of participants will be asked to provide the results of analyses performed in the routine clinical setting related to the participant's general health and the administration of velmanase alfa.

Additional data will be extracted from other observational sponsored studies/registries, compassionate use programs, investigator-initiated studies (IIS), and published case reports (presented in the literature) if existing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with the provision of informed consent from their legal guardians (LAR)
* Have a confirmed diagnosis of alpha mannosidosis
* Have initiated treatment with velmanase alfa between birth to at least six weeks before turning 3 years of age
* Have information on the disease marker GlcNAc(Man)2 obtained:

before velmanase treatment initiation (ideally max 6 month before), and at least one post-treatment sample, collected following at least six weeks of treatment.

- Participants treated with Lamzede, 1 mg/kg body weight, via weekly intravenous infusions.

Exclusion Criteria:

Participants who have undergone prior hematopoietic stem cell transplantation (HSCT) or other investigational therapies for treating alfa mannosidosis (supportive treatments acceptable).

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Paediatric patients with a confirmed diagnosis of alpha mannosidosis via MAN2B1 genetic testing and/or alpha-mannosidase activity in leukocytes or fibroblasts < 10% of normal activity, with data for at least one pre- and one post-Lamzede treatment sample obtained when < 3 YOA, after at least 6 weeks of treatment (primary analyses).
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamic Response to velmanase alfa | 52 weeks of treatment
  Change (absolute and relative) of GlcNAc(Man)2 level from pre-velmanase alfa treatment baseline in blood

OTHER OUTCOMES:
Development of anti drug antibody to velmanase alfa | 52 weeks of treatment
  Assessment of the impact of anti drug antibody on pharmacodinamic
Treatment-emergent adverse events | 52 weeks
  Number of undesirable events not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the treatment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Nicklaus Children's Hospital, Miami, Florida
  - Greenwood Genetic Center, Greenwood, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Chiesi site web study information — https://www.chiesiclinicalstudies.com/trials/CLI-LMZYMAA2-04